CLINICAL TRIAL: NCT06637085
Title: Acu Tens Versus Low Level Laser on Autonomic and Heamodynamic Stability After Open Heart Surgeries.
Brief Title: Acu Tens Versus Low Level Laser After Open Heart Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, haidy mustufa elmessallamy, assisstanr lecture at faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: p.T.REC/012/003894
Record Dates: First submitted 2024-05-01; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Heart Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- LLLT group (Experimental): The LLLT group consist of (20) patients, who will receive the vagus nerve stimulation through LLLT from the first day postoperative until the seventh day, in addition to routine physiotherapy program
  Interventions: Device: LLLT; Other: traditional physical therapy
- ACU tens group (Experimental): The acu tense group consist of (20) patients, who will receive the acu tens on (pc6) point from the first day postoperative until the seventh day, in addition to routine physiotherapy program
  Interventions: Other: traditional physical therapy; Device: ACU TENSE
- control group (Active Comparator): The control group consist of (20) patients, who will receive only routine physiotherapy program (phase I cardiac rehabilitation, breathing exercises, modified postural drainage, percussion and vibration)
  Interventions: Other: traditional physical therapy

INTERVENTIONS:
Device: LLLT — low level laser therapy Probe laser device: (Laserklasse2M, EN60825-1, +A2:2002, W.L= 635-670nm, P<6mW, German):low level laser therapy It will be used to stimulate vagus nerve .
  Arms: LLLT group
Other: traditional physical therapy — traditional physical therapy include (phase I cardiac rehabilitation, breathing exercises, modified postural drainage, percussion and vibration)
Device: ACU TENSE — Acu-TENS device (Digital TENS, EAF20, JERF20BD0604, add manufacturing country): It will be used to stimulate vagus nerve throug h the acupoint PC6 .
  Arms: ACU tens group

SUMMARY:
Increase in heart rate (HR) is a normal sympathetic response to body trauma and a common consequence of major surgical procedures,A high resting HR is associated with increased myocardial work that may be detrimental to patients with a marginal myocardial oxygen supply,the aim of this study is To compare between the effects of Acu TENS and low level laser therapy on autonomic and hemodynamic instability after open heart surgery.

DETAILED DESCRIPTION:
Autonomic function reached lowest values 3-6 days after coronary artery by pass graft (CABG) and could take up to 60 days to return to pre-surgery values (pedro et al., 2005).

Alterations in pulse may provide a first indication that a patient is developing hemodynamic instability. While many factors may influence the pulse rate, including fever, exercise, medications, and thyroid hormone status, a high pulse rate is often a sign of high levels of endogenous catecholamines, blood loss or dehydration (Jonathan ,2009.) Hemodynamically unstable patients don't have enough pressure in the circulatory system to keep blood flowing reliably to all the various parts of the body where it needs to be at the same time.

Vagus nerve stimulation (VNS) can increase HRV and reduce sympathetic nerve outflow, which is desirable in conditions characterized by enhanced sympathetic nerve activity .

Application of Acu-TENS over acu-point PC6 facilitated a faster return of resting HR to preoperative levels, maintained BP during the acute postoperative period and enhanced a quicker return of rate pressure product (RPP), in patients after acute cardiac surgery .

Faster return of the raised resting HR to preoperative levels in Acu-TENS application was possibly due to induced vagal stimulation and/or inhibition of sympathetic neural activity through the acu-points PC6 .

Low level laser therapy (LLLT) is a non-invasive and safe method, to recover parasympathetic/sympathetic nervous system balance .

this study show the differences between the effect of Acu TENS and low level laser therapy on autonomic and hemodynamic instability after open heart surgery

ELIGIBILITY:
Inclusion Criteria:

* 1- 60 patients from both sexes . 2- undergo cardiac surgery through a median sternotomy. 3- age will be ranged from 45-65 years old. 4-Body mass index from 25 to 29.9 kg/m25-

Exclusion Criteria:

* 1- Previous thoracic surgery. 2- Emergency or urgent cardiac surgery. 3- hypoxemia with partial pressure of oxygen in arterial blood <60 mmHg. 4- Renal insufficiency with serum creatinine ≤1.8 mg/dl after surgery. 5- Other medical conditions such as uncontrolled diabetes, and hypertension . 6- Patients who are unable to follow verbal instructions.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-11-05 (Actual); Study Completion 2024-02-03 (Actual)

PRIMARY OUTCOMES:
heartrate variability. | heart rate variability parameters recorded for 24 hours 1st day post operative and at the last day before discharge from hospital for each group. before discharge from hospital .
  SDANN Standard deviation of the averages of RR intervals in all 50minute segments of a 24-hour recording.rMSSD Square root of the mean of the squares of differences between adjacent RR intervals

SECONDARY OUTCOMES:
Atrial fibrillation | AF recorded in 24 hours 1st day post operative and at the last day before discharge from hospital for each group.
  Atrial fibrillation occurs in 10% to 65% of patients after cardiac surgery, usually on the second or third postoperative day. Postoperative atrial fibrillation is associated with increased morbidity and mortality and longer, more expensive hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: zeinab helmy, professor, Study Director — Cairo University
Locations (1):
- Kasr Ainy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chandler HK, Kirsch R. Management of the Low Cardiac Output Syndrome Following Surgery for Congenital Heart Disease. Curr Cardiol Rev. 2016;12(2):107-11. doi: 10.2174/1573403x12666151119164647. PMID 26585039
- [Background] Demirel S, Akkaya V, Oflaz H, Tukek T, Erk O. Heart rate variability after coronary artery bypass graft surgery: a prospective 3-year follow-up study. Ann Noninvasive Electrocardiol. 2002 Jul;7(3):247-50. doi: 10.1111/j.1542-474x.2002.tb00171.x. PMID 12167187
- [Background] Syuu Y, Matsubara H, Hosogi S, Suga H. Pressor effect of electroacupuncture on hemorrhagic hypotension. Am J Physiol Regul Integr Comp Physiol. 2003 Dec;285(6):R1446-52. doi: 10.1152/ajpregu.00243.2003. Epub 2003 Jul 31. PMID 12893654
- See also: Related Info — https://scholar.google.com/scholar?hl=ar&as_sdt=0%2C5&q=https%3A%2F%2Fwww.ingentaconnect.com%2Fcontent%2Fben%2Fccr%2F2016%2F00000012%2F00000002%2Fart00007&btnG=
- See also: Related Info — https://scholar.google.com/scholar?hl=ar&as_sdt=0%2C5&q=https%3A%2F%2Fonlinelibrary.wiley.com%2Fdoi%2Fabs%2F10.1111%2Fj.1542-474X.2002.tb00171.x&btnG=
- See also: Related Info — https://scholar.google.com/scholar?hl=ar&as_sdt=0%2C5&q=http%3A%2F%2Fhttps%3A%2F%2Fonlinelibrary.wiley.com%2Fdoi%2Fabs%2F10.1111
- See also: Related Info — https://scholar.google.com/scholar?hl=ar&as_sdt=0%2C5&q=http%3A%2F%2Fhttps%3A%2F%2Fwww.sciencedirect.com%2Fscience%2Farticle%2Fpii%2FS1935861X14002605&btnG=